CLINICAL TRIAL: NCT02720302
Title: Treatment of Overweight in Children on Distance. A Comparison Between Consultations on the Hospital With Video-Consultations on Distance
Brief Title: Treatment of Overweight in Children on Distance
Acronym: TeleSOFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Carl-Erik Flodmark, Docent, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/141
Record Dates: First submitted 2015-11-23; First posted 2016-03-25 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Overweight
Keywords: Overweight; Children; Treatment; Prevention; Lifestyle intervention
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOFT (Experimental): All Children have their first and their last consultation at The Child Obesity Unit.
  The investigators use Standardized Obesity Family Therapy "SOFT" as described by Nowicka & Flodmark (1-3). The intervention use psychological techniques developed in systemic family therapy applied on advice regarding exercise and diet as well as behavioural Life style Changes.
  At each consultation with the overweight child and his/her biological parents there are two therapists present.
  Interventions: Behavioral: SOFT
- TeleSOFT (Experimental): The same method Lifestyle intervention "SOFT" is used. The only difference is that the communication in the second, third (and fourth) visit is made by use of video on distance. The investigators use Standardized Obesity Family Therapy "SOFT" as described by Nowicka & Flodmark (1-3).
  Interventions: Behavioral: TeleSOFT

INTERVENTIONS:
Behavioral: SOFT — SOFT is based on systemic and solution-focused theories to change lifestyle and has shown positive effects on children with respect to the degree of obesity, physical fitness, self-esteem and family functioning.
  Arms: SOFT
Behavioral: TeleSOFT — The therapists communicate with the overweight child and his/her family by the SOFT method on distance by use of video.
  Arms: TeleSOFT

SUMMARY:
The present study is a public health project with the aim to treat overweight in children 9-11 years of age. After the first consultation the children are randomized to either continue the treatment at The Child Obesity Clinic, Child Department or to have the following 2-3 consultations on distance with Lync. Last visit for all children is on the Child Obesity Clinic after approximately 12 months. Follow up after at least 1 years will be performed.

DETAILED DESCRIPTION:
This superiority study is a randomized trial with two independent treatment arms. The target for the enrollment is 50% in each of the two treatment groups.

With 60 patients in each group, the study has 80% statistical power at 5% significance level to detect an average difference between the treatment groups in the intra-individual change in the BMI Z-score that is 0.51 x the standard deviation in the intra-individual change. Previous data from the investigators own group suggest that a reasonable estimate of the standard deviation in the intra-individual change in the BMI Z-score following intervention is 0.42. Thus, the study has 80% statistical power at 5% significance level to detect a difference in the intra-individual change in the BMI Z-score that is 0.51 x 0.42 = 0.21 on average. The study will with the present funding end its follow up in June 2017.

ELIGIBILITY:
Inclusion Criteria:

- Children with overweight and not obese according to the definitions developed by Cole et al (4). It implies that we include children with the following age specific BMI Inclusion criteria

* 9 years = AGE < 9 years, 6 months AND 19,0< BMI<23,0
* 9 years, 6 months => AGE < 10 Years AND 19,5 <BMI<23,5
* 10 years = AGE < 10 years, 6 months AND 20,0<BMI<24,0
* 10 years, 6 months=>AGE< 11 years AND 20,5<BMI<24,5
* 11 years = AGE < 11 years, 6 months AND 21,0<BMI<25,5
* 11 years, 6 months =>AGE<12 years AND 21,5<BMI<25,5

Exclusion Criteria:

* Children and his/her parents not able to communicate in Swedish.
* Children with monogenic obesity
* Present less than 80% at school in the latest school year.
* No foster care for the child or his/her brothers or sisters

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index standard deviation score (BMI Z-score) during treatment of overweight | Change from Baseline in body weight at an average of 12 months
  Body weight measured by Tanita device

SECONDARY OUTCOMES:
Change in fat percent measured by TANITA | Change from Baseline in fat percent at an average of 12 months
  TANITA measures fat percent via bioimpedance
Change in fat distribution measured by abdominal height (F-indicator) | Change from Baseline in fat distribution at an average of 12 months
  F-indicator uses a laser beam to measure the abdominal height
Change in fat distribution measured by waist circumference | Change from Baseline in waist circumference at an average of 12 months
  Measured using a measurement tape
Change in KIDSCREEN-index | Change from Baseline in Kidscreen index at an average of 12 months
  Use a validated questionnaire
Change in physical activity measured by Moves application to smartphone | Change from Baseline in physical activity at an average of 2, 4, 6, 8, 12 months
  Measured through an app on a smart phone.
Change child's metabolic health (Blood pressure) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (LDL-cholesterol) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (HDL-cholesterol) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (triglycerides) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (HbA1c) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (F-blood glucose) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (f-insulin) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (ccK-18) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change child's metabolic health (ALAT) | Change from Baseline in metabolic health at an average of 12 months
  Standardized laboratory tests will be performed
Change in dietary habits | Change from Baseline in dietary habits at an average of 12 months
  Normal procedure at The Child Obesity Unit using a questionnaire
Change in Outcome Rating Scale and Session Rating Scale | Change from Baseline in Outcome Rating Scale at an average of 2, 4, 6, 8, 12 months
  Measured psychological Health in general by four questions combined to a general score on a Visual analogue scale
Change in Session Rating Scale | Change from Baseline in Session Rating scale at an average of 2, 4, 6, 8, 12 months
  Measured assessment of the consultation by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Agardh, Professor, Study Chair — Skane University Hospital
Locations (1):
- Barnmedicin, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowicka P, Pietrobelli A, Flodmark CE. Low-intensity family therapy intervention is useful in a clinical setting to treat obese and extremely obese children. Int J Pediatr Obes. 2007;2(4):211-7. doi: 10.1080/17477160701379810. PMID 17852553
- [Background] Flodmark CE, Ohlsson T, Ryden O, Sveger T. Prevention of progression to severe obesity in a group of obese schoolchildren treated with family therapy. Pediatrics. 1993 May;91(5):880-4. PMID 8474806
- [Background] Nowicka P, Flodmark CE. Family therapy as a model for treating childhood obesity: useful tools for clinicians. Clin Child Psychol Psychiatry. 2011 Jan;16(1):129-45. doi: 10.1177/1359104509355020. Epub 2010 Jul 22. PMID 20650975
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032